CLINICAL TRIAL: NCT05220293
Title: The Effect of Betamethasone Dipropionate on Patients With Eosinophilic Chronic Rhinosinusitis
Brief Title: Treatment of Eosinophilic Chronic Rhinosinusitis Utilizing Betamethasone Dipropionate Nasal Cream
Acronym: OT-007
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Single site study OT-007 re-opened as multi-site OT-007B study
Sponsor: Oticara Australia PTY LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OT-007
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Chronic Rhinosinusitis (Diagnosis)
Keywords: eosinophilic Chronic Rhinosinusitis
MeSH Terms: conditions — Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Betamethasone Dipropionate Nasal Cream 0.0644% Treatment (Experimental): Betamethasone Dipropionate Nasal Cream 0.0644% is applied topically to the inflamed tissue of the sinus using a pre-filled syringe and applicator under the guidance of an endoscope. Up to 5g on each side of the sinus (10g in total).
  Interventions: Drug: Betamethasone Dipropionate Nasal Cream 0.0644%; Device: Pre-filled syringe and applicator device

INTERVENTIONS:
Drug: Betamethasone Dipropionate Nasal Cream 0.0644% — Betamethasone Dipropionate Nasal Cream 0.0644%, up to 5g per sinus.
Device: Pre-filled syringe and applicator device — Cream is pre-filled to a syringe and applicator device to facilitate the topical application direct to the sinus under endoscopic guidance.

SUMMARY:
This is an open-label, single dose, pilot study, to assess the efficacy and safety of Betamethasone Dipropionate Nasal Cream 0.0644% (equivalent to 0.05% Betamethasone) for the treatment of eosinophilic Chronic Rhinosinusitis (eCRS).

DETAILED DESCRIPTION:
In this open-label study, a single dose of the corticosteroid Betamethasone Dipropionate Nasal Cream 0.0644% (equivalent to 0.05% Betamethasone) will be administered under endoscopic guidance to the sinus mucosa of post-FESS patients whose eCRS condition is suboptimal under the current standard of care. The safety and benefits of this treatment will be monitored by patient-reported symptoms and visualization of the sinus mucosa.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a clinically confirmed diagnosis of eCRS by a ENT undergoing maximal medical therapy as part of their standard of care.
* Having undergone functional endoscopic sinus surgery at least 6 months prior to enrolment.
* Participants with an endoscopic bilateral nasal polyp score of ≤5 out of a maximum score of 8
* Score > 2 on disease severity visual analogue scale (VAS)
* A minimum body weight >=40 kilograms (kg) at screening visit
* Gender: Male or female (females of childbearing potential must use adequate birth control methods and not plan to get pregnant during the course of the study).
* Informed consent: Willingness to give written informed consent and willingness to participate to and comply with the study.
* Age ≥18 but <80 years.

Exclusion Criteria:

* Subjects with known hypersensitivity or contraindications to Betamethasone Dipropionate, corticosteroids or topical anaesthesia.
* Subjects with sino-nasal abnormalities, disease or implanted devices that prevent application of the therapy.
* Previous enrolment in this study.
* Subjects currently required systemic corticosteroid use or receiving biologic therapy as part of their disease management plan or who meet the PBS criteria for severe lower airway disease.
* Subjects with history or current glaucoma or cataract or if they have abnormal IOP at screening or pre-treatment (abnormal IOP is defined as greater than 21 mm Hg).
* Subjects with other conditions that could lead to elevated eosinophils such as Hypereosinophilic Syndromes, including Churg-Strauss Syndrome, or Eosinophilic Esophagitis.
* Subjects with acute sinusitis.
* Subjects with known immunodeficiency.
* Subjects with Diabetes (Type 1).
* Subjects with cystic fibrosis.
* Pregnant subjects or subjects currently lactating as the effect on human pregnancy is unknown.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-02-23 (Actual); Primary Completion 2023-12-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Change in 4 cardinal symptoms score (4CSS) from Baseline to Week 3. | Baseline to Week 3
  Participants score their 4-Cardinal Symptom score (4CSS) daily on a Likert scale of 0-5; where 0= no problem - 5= problem as bad as can be, higher scores indicate higher severity of symptoms.
Change in Visual Analogue Scale (VAS) (0-10) evaluating global disease severity score from Baseline to Week 3. | Baseline to Week 3
  Participants score their global disease severity assessment daily on a Visual Analogue Scale (VAS) (0-10), higher score indicating greater disease severity.
Change in SNOT-22 Score from Baseline to Week 3. | Baseline to Week 3
  Participants complete the SNOT-22 questionnaire at Baseline and Week 3,analysis will focus on the nasal and ear/facial subdomains. Higher scores indicate greater severity.
Change in Modified Lund Mackay Postoperative Endoscopy Score from Baseline to Week 3. | Baseline to Week 3
  Change in Modified Lund Mackay Postoperative Endoscopy Score is evaluated by experienced ENT at Baseline to Week 3.
Overall Patient Global Impression of Change at Week 3. | Week 3
  Patient Global Impression of Change (recorded on a Likert scale 1-7, where 1= very much improved - 7= very much worse) will be completed by the participant at Week 3.

SECONDARY OUTCOMES:
BMDP Cream retention time on the sinus | Treatment visit to Week 3
  Visual inspection of cream retention time on the sinus via endoscope.
To assess the safety of one application of BMDP CREAM onto the sinus | Treatment visit to Week 3
  Adverse event and intraocular pressure monitoring

CONTACTS AND LOCATIONS:
Overall Officials: Oticara Clinical, Study Director — Oticara Australia PTY LTD
Locations (1):
- Oticara Clinical Trial Site, Sydney, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.